CLINICAL TRIAL: NCT06110143
Title: The Prevention of Adverse Pregnancy Outcomes by Periodontal Treatment (PROBE) Intervention Study
Brief Title: Oral Health and Adverse Pregnancy Complications
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Bispebjerg and Frederiksberg (Other)
Responsible Party: Principal Investigator, Karoline Winckler, Phd, postdoc, University Hospital Bispebjerg and Frederiksberg
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H-20083249
Record Dates: First submitted 2023-10-25; First posted 2023-10-31 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Periodontal Diseases; Pregnancy Complications; Pregnancy Preterm; Gestational Diabetes; Preeclampsia; Inflammation
MeSH Terms: conditions — Periodontal Diseases; Pregnancy Complications; Diabetes, Gestational; Pre-Eclampsia; Inflammation | interventions — Periodontal Index

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- PrePROBE (Other): Periodontal treament during pregnancy
  Interventions: Other: Periodontal treatment
- PostPROBE (Other): Peridontal treatment postpartum
  Interventions: Other: Periodontal treatment

INTERVENTIONS:
Other: Periodontal treatment — Periodontal treatment

SUMMARY:
Pregnant women are susceptible to develop periodontitis, but these oral health changes related to pregnancy are often neglected. Periodontitis is accompanied by a low-grade systemic inflammation and can be harmful to the general health of the woman, contribute to pre-term birth and adversely influence the future health and metabolism of the offspring. Despite this, studies indicate that 40% of Danish women in childbearing age do not visit a dentist regularly. The PROBE controlled intervention study will investigate the beneficial effect of treatment of periodontal disease during pregnancy on fetal growth, preterm delivery and birth weight.

DETAILED DESCRIPTION:
Periodontitis is one of the most common and chronic inflammatory oral conditions reaching approximately 20 - 60 % of the global population. The disease is characterized as a set of inflammatory conditions affecting the tissues surrounding the teeth. In the early stages, called gingivitis, where the disease is still reversible, the gums can become swollen, red and may bleed. Later in the disease development, periodontitis will progress into a more chronic condition. If untreated, periodontitis can cause tooth loss resulting in several complications including impaired speech, low self-esteem and reduced ability to eat freely and accumulating evidence has now linked periodontitis to a wide range of common medical conditions.

Pregnant women are susceptible to develop periodontitis due to hormonal changes leading to increased blood flow, plaque retention and risk of gingival infection, that may progress to periodontitis if persisting untreated. The prevalence of periodontitis in pregnancy has not been systematically assessed and varies significantly across studies with a range of 0 % -61 %. This large variation might be attributed to the diverse definitions of periodontitis. Still, optimal oral health care during pregnancy is often neglected and numbers from the Danish Dental Association indicate that 40% of Danish women in childbearing age do not visit a dentist regularly. Apart from the oral consequences resulting from periodontitis the condition is accompanied by a low-grade systemic inflammation. The systemic inflammation caused by periodontitis during pregnancy may have consequences beyond the oral cavity. Systematic reviews have shown that women with periodontitis can adversely influence the future health and metabolism of the offspring by an increased risk of preterm birth (< 37 weeks gestation) and delivering babies with low-birth-weight (< 2.5 kg). However, the biological mechanism underlying the link between periodontitis and adverse pregnancy outcomes is not fully known.

Early prevention of periodontal disease among pregnant women may have beneficial effects for both the mother and child. Providing periodontal treatment for pregnant women might reduce the risk of preterm birth, low birthweight as well as risk markers for pre-eclampsia and gestational disease. The idea and ambition of the prevention of adverse pregnancy outcomes by periodontal treatment' (PROBE) controlled intervention study is to investigate the beneficial effect of treatment of periodontal disease during pregnancy on fetal growth, preterm delivery and birth weight. Firstly, by investigating the prevalence of periodontitis among pregnant women. Secondly to prevent development of periodontal disease and the related systemic inflammation during pregnancy by intervening with periodontal treatment to reduce the risk of pregnancy and birth related outcomes. Reducing the development of these outcomes are expected to limit the risk of later development of metabolic disturbances in the offspring. Another implication of minimizing the prevalence of periodontitis is the potential reduction in other chronic diseases that periodontitis has been linked to, e.g. diabetes, cardiovascular disease and Alzheimer's.

If the key findings from the PROBE study are positive, the main message will be that oral hygiene and prevention of periodontitis during pregnancy are important and that treatment and regular visits to a dentist needs priority during pregnancy. Offering free dental care during pregnancy in Denmark would in the already established clinics be an easy implementable strategy to reduce adverse pregnancy and birth related outcomes. There will be economic costs related to providing free dental care, but the long-term beneficial effects both for the women and children as well as for society are expected to be significant and may exceed the costs of the intervention.

The overall aims of the study are to:

1. Investigate the prevalence of periodontitis in pregnant women and whether periodontal treatment during pregnancy can improve the periodontal condition (less pocket depth, bleeding on probing and attachment loss) and reduce the systemic inflammation.
2. Investigate whether periodontal treatment contributes to a reduced risk of preterm birth, low birthweight and lower risk markers of preeclampsia and gestational diabetes (blood pressure and hemoglobin A1c (HbA1c)).

The PROBE study is a controlled intervention study, where approximately 1200 pregnant women will be recruited from either Holbæk Hospital or Nykøbing Falster Hospital in Region Zealand in Denmark during their nuchal fold scan in gestation week 11-14 following a periodontal screening visit at the study dentist. During the nuchal fold scan, the secretaries will hand out documents to all pregnant women attending the scan. Inclusion criteria are pregnant women who speaks and understand Danish and is diagnosed with periodontitis by the study dentist. Exclusion criteria are pregnant women without periodontitis. The secretaries at Holbæk and Nykøbing Falster Hospitals will coordinate the recruitment and inclusion of participants for the study. Information on eligible participants will be given to the research coordinator and the research dentist by the secretaries. It is expected that 50 % of the screened population will be diagnosed with periodontitis and suitable for inclusion. The intervention group of approximately 300 pregnant women with periodontitis, receives periodontal treatment during pregnancy, and the control group of approximately 300 pregnant women with periodontitis, receives periodontal treatment after giving birth. The method and data collection activities are the same for both the intervention and the control group, except for the time of the periodontal treatments that are performed during pregnancy and after birth. The time period for the periodontal treatments will be the same for each group, approximately 20 weeks, and each included participant can receive up to 5 periodontal treatments. Recruitment of pregnant women with periodontitis will last over a period of 18 months for the intervention group and additional 18 months for the control group.

Demographic information, qualitative questionnaires related to diet, smoking status, physical activity, family status, socio economic status and oral health care and dental habits will be collected at baseline (week 11-13 of gestation) and at week 35 of gestation through online questionnaires. Two months and six months post-partum two additional qualitative questionnairea regarding growth of the baby, and questions about the partner, oral health and dental habits will be send through online questionnaire.

Regional dental clinics in Region Zealand have been approached in relation to possibilities of providing available clinics. The clinics have responded positively and are willing to provide the clinics also outside normal opening hours, which would facilitate potential implementation of the project afterwards.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women who are planned to give birth at either Holbaek or Nykoebing Falster hospital
* Pregnant women diagnosed with periodontitis (stage I-III) by the study dentist

Exclusion Criteria:

* Pregnant women without peridontitis
* Pregnant women with less than 20 healthy teeths
* Pregnant women with peridontitis and currently receiving treatment for peridontitis
* Pregnant women with peridontitis stage IV

Ages: 16 Years to 48 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 600 (Estimated)
Dates: Start 2021-11-13 (Actual); Primary Completion 2025-11 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Prevalence of preterm birth | 18 months
  Defined as any birth before 37 completed weeks of gestation
Prevalence of low birthweight | 18 months
  Defined as a birth weight of less than 2500 gram
Increased risk markers for preeclampsia | 18 months
  Defined as hypertension and proteinuria
Prevalence of gestational diabetes | 18 months
  Defined as glucose intolerance

CONTACTS AND LOCATIONS:
Overall Officials: Berit Lilienthal Heitmann, Professor, Principal Investigator — University Hospital Bispebjerg and Frederiksberg
Locations (3):
- Denmark (3):
  - Holbaek Hospital, Holbæk, Holbaek
  - Holbæk Hospital, Holbæk, Holbaek
  - Nykøbing Falster Hospital, Nykøbing Falster, Nykøbing Falster

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Winckler K, Bukkehave KH, Tarnow L, Iversen PB, Damgaard C, Ditlev SB, Kofoed-Enevoldsen A, Fischer HM, Dueholm SCH, Lauenborg J, Trier C, Heitmann BL. The prevention of adverse pregnancy outcomes by periodontal treatment during pregnancy (PROBE) intervention study-A controlled intervention study: Protocol paper. PLoS One. 2024 May 13;19(5):e0302010. doi: 10.1371/journal.pone.0302010. eCollection 2024. PMID 38739615